CLINICAL TRIAL: NCT05038306
Title: Chinese Medicine WT for Elevating IGF-1 of Patients With Spinocerebellar Ataxia Type 3 - Pilot Study
Brief Title: Chinese Medicine WT for Spinocerebellar Ataxia Type 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Chiu Chung Min, Adjunct Physician, Changhua Christian Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200703
Record Dates: First submitted 2021-05-27; First posted 2021-09-09 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Ataxia, Spinocerebellar; Insulin-Like Growth Factor I; Medicine, Chinese Traditional
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese Medicine (Active Comparator)
  Interventions: Drug: Chinese medicine WT
- Placebo (Placebo Comparator)
  Interventions: Drug: Chinese medicine WT

INTERVENTIONS:
Drug: Chinese medicine WT — The Chinese medicine WT is thought to be neurotrophic, and its major constituent may benefit IGF-1 in animal studies, or certain healthy human group. WT is safe in clinical use in Asia.

SUMMARY:
Spinocerebellar ataxia type 3 (SCA3) is one of autosomal dominant hereditary ataxias. Standing imbalance, unsteady gait, dysmetria, fatigue, and depression would occur gradually. There are no effective treatment or palliative methods for patients in the present days. However, low-dose growth hormone, or its downstream product, insulin-like growth factor I (IGF-1), may deter the progress of SCA3 in transgenic mice. The main bioactive constituent among the Chinese medicine WT possesses neuroprotective function against glutamate-induced toxicity, which is one major pathology of SCA3. It promotes neurogenesis, and increases the protein expression of IGF-1 in ischemic brains of rats. Thus, we designed a randomized, double-blind trial for patients with SCA3, if WT is a possible neuroprotective medicine.

All the subjects will be recruited from Changhua Christian Hospital. Diagnosis is confirmed by gene test and magnetic resonance image by a neurologist. They will be assigned in random and double blind, prescribed with 3 grams concentrated powder of WT or placebo, twice a day, for 12 weeks. After the washout period of 4 weeks, there will be a crossover of placebo or WT for another 12 weeks. After that, another 4-week rest will be followed by the end of trial. Check items in five check points include: 1. Blood examination (serum IGF-1, Neurofilament light chain, mitochondria copy number, 8_OHdG, delta-Ct), 2.Neurological exam (Scale for the Assessment and Rating of Ataxia), 3. Questionnaires (Modified Fatigue Impact Scale, Epworth Sleepiness Scale), 4. Handgrip strength test (which is correlated to IGF-1 value in elderly), and 5. serum metabolites, . All the data will be disclosed after the end of trial. Paired-T test or Wilcoxon Ranked Sign Test will be operated in SPSS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as Spinocerebellar Ataxia type 3

Exclusion Criteria:

* 1. using other Chinese medicine or herbal medicine 2. allergic to Chinese medicine or herbal medicine 3. pregnancy or breast feeding 4. with other major diseases, such as cancer, stroke, heart failure, or renal failure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Insulin-like Growth Factor 1 at week 12, or from week 16 to week 28 | baseline and 12 weeks, or 16 weeks and 28 weeks, 32 weeks
  Insulin-like growth factor I is appropriate to observe the change for a period instead of the absolute value.
Change from baseline in Neurofilament light Chain at week 12, or from week 16 to week 28 | baseline and 12 weeks, or 16 weeks and 28 weeks, 32 weeks
  Neurofilament light Chain is appropriate to observe the change for a period instead of the absolute value

SECONDARY OUTCOMES:
Change from baseline in scale for the assessment and rating of ataxia(SARA) at week 12, or from week 16 to week 28 | baseline and 12 weeks, or 16 weeks and 28 weeks
  scores of SARA are from 0 to 40, with higher scores means worse outcome
Change from baseline in Modified Fatigue Impact Scale (MFIS) at week 12, or from week 16 to week 28 | baseline and 12 weeks, or 16 weeks and 28 weeks
  scores of MFIS are from 0 to 84, with higher scores means worse outcome
Change from baseline in Epworth Sleepiness Scale (ESS) at week 12, or from week16 to week 28 | baseline and 12 weeks, or 16 weeks and 28 weeks
  scores of ESS are from 0 to 24, with higher scores means worse outcome
Change from baseline in Hand-grip strength test (HST) at week 12, or from week16 to week 28 | baseline and 12 weeks, or 16 weeks and 28 weeks
  HST is appropriate to observe the change for a period instead of the absolute value
Change from baseline in mitochondria DNA (mtDNA) at week 12, or from week16 to week 28 | baseline and 12 weeks, or 16 weeks and 28 weeks
  mitochondrial DNA HST is appropriate to observe the change for a period instead of the absolute value
Change from baseline in 8_OHdG at week 12, or from week16 to week 28 | baseline and 12 weeks, or 16 weeks and 28 weeks
  8_OHdG is appropriate to observe the change for a period instead of the absolute value
Change from baseline in △Ct at week 12, or from week16 to week 28 | baseline and 12 weeks, or 16 weeks and 28 weeks
  △Ct is appropriate to observe the change for a period instead of the absolute value
Change from baseline in serum metabolites at week 12, or from week 16 to week 28 | baseline and 12 weeks, or 16 weeks and 28 weeks
  serum metabolites is appropriate to observe the change for a period instead of the absolute value. Till now, there was no sufficient data about the metabolites of Chinese WT, so we would like to measure the difference of metabolites before and after taking the Chinese medicine WT.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No